CLINICAL TRIAL: NCT01319825
Title: Open Label Study of Milnacipran in the Preventive Treatment of Episodic Migraine With and Without Aura and Chronic Migraine.
Brief Title: Preventive Treatment of Episodic and Chronic Migraine
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: California Medical Clinic for Headache (Other)
Responsible Party: David Kudrow, M.D., California Medical Clinic for Headache
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SAV-MD-26
Record Dates: First submitted 2011-03-18; First posted 2011-03-22 (Estimated); Last update posted 2011-03-22 (Estimated); Status verified 2011-03

CONDITIONS: Migraine With Aura; Migraine Without Aura; Chronic Migraine
MeSH Terms: conditions — Migraine with Aura; Migraine without Aura | interventions — Milnacipran

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: milnacipran — 100 mg and 200 mg orally daily for a total of 4 months including a one month titration period.

SUMMARY:
This is an open label pilot study to determine whether milnacipran can reduce headache frequency in episodic and chronic migraine sufferers.

DETAILED DESCRIPTION:
Patients with episodic migraine with and/or without aura and chronic migraine will be treated with 100 or 200 mg of milnacipran for a total of 4 months including a one month titration phase and a 3 month maintenance phase. Baseline (pre-treatment) and end-of-maintenance phase headache frequencies will be recorded. There is no placebo treatment in this study. In addition to headache frequencies, other parameters being measured include safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Migraine with or without aura or chronic migraine.
* Subject age 18 to 70.
* At least 2 migraine attacks per month.
* Willing ang able to give written informed consent.
* Willing and able to complete the entire course of the study and to comply with study instructions.
* Willing to taper and discontinue their current preventive medications.

Exclusion Criteria:

* Subject is pregnant, lactating or planning a pregnancy in the next year.
* Subject is female of child-bearing potential and not taking adequate forms of birth control.
* Significant medical or psychiatric disease or abnormal laboratory data that would preclude entry into this study.
* Previous failure of four or more adequate trials of preventive medication.
* Currently on any form of antidepressant for depression and not able to discontinue.
* Currently demonstrating medication overuse headache.
* Currently has uncontrolled narrow angle glaucoma.
* Currently taking monoamine oxidase inhibitors.
* Subject has a history of seizures.
* Participation in an investigational drug study within the last 30 days or 5 half-lives, whichever is longer.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2011-04; Primary Completion 2012-05 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Reduction in number of all headache days per month in the last month of stable dosing, compared to baseline | 4 months

SECONDARY OUTCOMES:
Reduction in number of migraine days per month in the last month of stable dosing compared to baseline. | 4 months
Improvement in headache index score | 4 months
  Headache index is defined by headache severity x headache duration.
Reduction in the number of days of headache related disability/impairment | 4 months
Tolerability | 4 months
  Assessment of adverse events
Use of rescue medications | 4 months
  To assess the continued need for acute headache treatments during the study period.
Quality of life measures | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: David B Kudrow, MD, Principal Investigator — California Medical Clinic for Headache
Locations (1):
- California Medical Clinic for Headache, Santa Monica, California, United States

REFERENCES:
- [Derived] Engel ER, Kudrow D, Rapoport AM. A prospective, open-label study of milnacipran in the prevention of headache in patients with episodic or chronic migraine. Neurol Sci. 2014 Mar;35(3):429-35. doi: 10.1007/s10072-013-1536-0. Epub 2013 Sep 13. PMID 24030685
- See also: California Medical Clinic for Headache — http://www.clinicaltrialsla.com